CLINICAL TRIAL: NCT05445973
Title: Real-Time Contrast-Enhanced Ultrasonography-CT/MRI Fusion Guidance for Percutaneous Radiofrequency Ablation of Inconspicuous, Small Liver Tumors
Brief Title: Added Value of Contrast-enhanced Ultrasonography for Percutaneous Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUNH 1811-136-989
Record Dates: First submitted 2022-06-17; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Radiofrequency Ablation; Ultrasonography; Liver Tumors
Keywords: Percutaneous Radiofrequency Ablation; Real-Time Contrast-Enhanced Ultrasonography; Small Liver Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real-Time Contrast-Enhanced Ultrasonography-CT/MRI Fusion Guidance (Experimental): To investigate whether CEUS-CT/MRI fusion imaging improved the visualization of small (≤ 3 cm) primary and secondary malignant liver tumors that were inconspicuous on B-mode US for percutaneous RFA.
  Interventions: Procedure: Percutaneous Radiofrequency Ablation

INTERVENTIONS:
Procedure: Percutaneous Radiofrequency Ablation — In brief, ablation was performed using a 200-W multichannel generator and a switching monopolar technique with separate clustered electrodes. Tumor targeting was done under the guidance of CEUS-CT/MRI FI, and the ablation procedure was monitored with US-FI. The ablation procedure was terminated when the operator expected to complete the ablation of the index tumor with a minimum 5-mm ablative margin on the US-FI images.

SUMMARY:
Contrast-enhanced ultrasonography (CEUS)-CT/MRI fusion imaging substantially improved the visibility of small tumors that were inconspicuous on both US and US-CT/MRI fusion imaging, contributing to successful percutaneous radiofrequency ablation.

DETAILED DESCRIPTION:
Percutaneous radiofrequency ablation (RFA) has been widely implemented as a curative treatment for liver malignancies. The overall survival post-RFA is comparable to that of surgical outcomes for small hepatocellular carcinomas (HCCs) (≤ 3 cm). US guidance for RFA is common in Asia because the real-time capability of US allows precise electrode placement. However, precisely targeting small liver malignancies with poor sonographic conspicuity in US-guided RFA is often challenging. To solve this problem, CEUS or real-time fusion imaging (FI) of US and CT/MRI have been used. Both approaches have been reported to improve the confidence for tumor localization in RFA for small HCCs with poor B-mode US visibility. However, when an index tumor is entirely invisible on B-mode US, neither method is ideal, especially for multiple-electrode RFA, due to inherent registration errors on FI or insonation-induced bubble destruction on CEUS with SonoVue. Therefore, there is a clinical need to compensate for the inherent registration errors of US-CT/MRI FI for inconspicuous tumors on both US and US-CT/MRI FI.

Recent studies reported that after adding CEUS using Sonazoid (GE Healthcare, Waukesha, WI, USA) or SonoVue to FI, 83.3% to 90% of target liver cancers that were initially difficult to visualize on FI became conspicuous, allowing them to be directly targeted for RFA. However, these studies had limitations, including a retrospective study design, a small sample size (< 30 inconspicuous tumors), or a short-term follow-up (< 1 year). Furthermore, no prospective study has explored the value of CEUS-CT/MRI FI, using both SonoVue and Sonazoid as contrast agents, for localizing index tumors and guiding RFA procedures in patients with inconspicuous tumors on B-mode US and reported its therapeutic impact on local tumor control.

Therefore, the present study investigated whether CEUS-CT/MRI FI improved the visibility of small (≤ 3 cm) primary and secondary liver tumors that were invisible or difficult to visualize on B-mode US for percutaneous RFA.

ELIGIBILITY:
Inclusion Criteria:

* inconspicuous or invisible index tumors for ablation on US
* tumor size ≤ 3 cm
* pathologic diagnosis of primary or secondary liver malignancy or imaging-based diagnosis of HCC according to the American Association for the Study of Liver Disease guidelines or viable HCC according to the Liver Imaging Reporting and Data System treatment response algorithm
* consideration of curative-intent RFA

Exclusion Criteria:

* well-visible tumors (visibility score of 3 or 4) on the planning B-mode US
* the absence of available data from multiphase CT or MRI performed in the 3-month pre-procedure period
* poor quality registration of US-CT/MRI fusion imaging and RFA planned with palliative intent
* contraindications for the conventional RFA procedure at the authors' institution, which are uncontrollable coagulopathy (platelet count < 50,000/μL or international standard ratio ≥ 1.6), a low level of cooperation, impracticality of sedation, portal vein thrombus, the tumor abutting the portal vein, or larger bile ducts than the segmental branches

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Local tumor progression rate | 12 months after the radiofrequency ablation
  Evaluate local tumor progression by follow-up computed tomography (CT) or magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Technical success rate of radiofrequency ablation using contrast-enhanced US-CT/MRI fusion image | Immediately after radiofrequency ablation
  The technical success of radiofrequency ablation is defined as complete ablation of tumor with safety margin and evaluated by immediate post-procedural computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DH, Lee JM. Recent Advances in the Image-Guided Tumor Ablation of Liver Malignancies: Radiofrequency Ablation with Multiple Electrodes, Real-Time Multimodality Fusion Imaging, and New Energy Sources. Korean J Radiol. 2018 Jul-Aug;19(4):545-559. doi: 10.3348/kjr.2018.19.4.545. Epub 2018 Jun 14. PMID 29962861
- [Background] Ahmed M, Solbiati L, Brace CL, Breen DJ, Callstrom MR, Charboneau JW, Chen MH, Choi BI, de Baere T, Dodd GD 3rd, Dupuy DE, Gervais DA, Gianfelice D, Gillams AR, Lee FT Jr, Leen E, Lencioni R, Littrup PJ, Livraghi T, Lu DS, McGahan JP, Meloni MF, Nikolic B, Pereira PL, Liang P, Rhim H, Rose SC, Salem R, Sofocleous CT, Solomon SB, Soulen MC, Tanaka M, Vogl TJ, Wood BJ, Goldberg SN; International Working Group on Image-Guided Tumor Ablation; Interventional Oncology Sans Frontieres Expert Panel; Technology Assessment Committee of the Society of Interventional Radiology; Standard of Practice Committee of the Cardiovascular and Interventional Radiological Society of Europe. Image-guided tumor ablation: standardization of terminology and reporting criteria--a 10-year update. J Vasc Interv Radiol. 2014 Nov;25(11):1691-705.e4. doi: 10.1016/j.jvir.2014.08.027. Epub 2014 Oct 23. PMID 25442132
- [Background] Feng K, Ma KS. Value of radiofrequency ablation in the treatment of hepatocellular carcinoma. World J Gastroenterol. 2014 May 28;20(20):5987-98. doi: 10.3748/wjg.v20.i20.5987. PMID 24876721
- [Background] Gao J, Wang SH, Ding XM, Sun WB, Li XL, Xin ZH, Ning CM, Guo SG. Radiofrequency ablation for single hepatocellular carcinoma 3 cm or less as first-line treatment. World J Gastroenterol. 2015 May 7;21(17):5287-94. doi: 10.3748/wjg.v21.i17.5287. PMID 25954102
- [Background] Lee DH, Kim JW, Lee JM, Kim JM, Lee MW, Rhim H, Hur YH, Suh KS. Laparoscopic Liver Resection versus Percutaneous Radiofrequency Ablation for Small Single Nodular Hepatocellular Carcinoma: Comparison of Treatment Outcomes. Liver Cancer. 2021 Feb;10(1):25-37. doi: 10.1159/000510909. Epub 2021 Jan 14. PMID 33708637
- [Background] Lee MW, Kang D, Lim HK, Cho J, Sinn DH, Kang TW, Song KD, Rhim H, Cha DI, Lu DSK. Updated 10-year outcomes of percutaneous radiofrequency ablation as first-line therapy for single hepatocellular carcinoma < 3 cm: emphasis on association of local tumor progression and overall survival. Eur Radiol. 2020 Apr;30(4):2391-2400. doi: 10.1007/s00330-019-06575-0. Epub 2020 Jan 3. PMID 31900708
- [Background] Dietrich CF, Nolsoe CP, Barr RG, Berzigotti A, Burns PN, Cantisani V, Chammas MC, Chaubal N, Choi BI, Clevert DA, Cui X, Dong Y, D'Onofrio M, Fowlkes JB, Gilja OH, Huang P, Ignee A, Jenssen C, Kono Y, Kudo M, Lassau N, Lee WJ, Lee JY, Liang P, Lim A, Lyshchik A, Meloni MF, Correas JM, Minami Y, Moriyasu F, Nicolau C, Piscaglia F, Saftoiu A, Sidhu PS, Sporea I, Torzilli G, Xie X, Zheng R. Guidelines and Good Clinical Practice Recommendations for Contrast-Enhanced Ultrasound (CEUS) in the Liver-Update 2020 WFUMB in Cooperation with EFSUMB, AFSUMB, AIUM, and FLAUS. Ultrasound Med Biol. 2020 Oct;46(10):2579-2604. doi: 10.1016/j.ultrasmedbio.2020.04.030. Epub 2020 Jul 24. PMID 32713788
- [Background] Mauri G, Cova L, De Beni S, Ierace T, Tondolo T, Cerri A, Goldberg SN, Solbiati L. Real-time US-CT/MRI image fusion for guidance of thermal ablation of liver tumors undetectable with US: results in 295 cases. Cardiovasc Intervent Radiol. 2015 Feb;38(1):143-51. doi: 10.1007/s00270-014-0897-y. Epub 2014 May 8. PMID 24806953
- [Background] Minami Y, Kudo M. Review of dynamic contrast-enhanced ultrasound guidance in ablation therapy for hepatocellular carcinoma. World J Gastroenterol. 2011 Dec 7;17(45):4952-9. doi: 10.3748/wjg.v17.i45.4952. PMID 22174544
- [Background] Francica G, Meloni MF, Riccardi L, de Sio I, Terracciano F, Caturelli E, Iadevaia MD, Amoruso A, Roselli P, Chiang J, Scaglione M, Pompili M. Ablation treatment of primary and secondary liver tumors under contrast-enhanced ultrasound guidance in field practice of interventional ultrasound centers. A multicenter study. Eur J Radiol. 2018 Aug;105:96-101. doi: 10.1016/j.ejrad.2018.05.030. Epub 2018 May 31. PMID 30017305
- [Derived] Lee Y, Yoon JH, Han S, Joo I, Lee JM. Contrast-enhanced ultrasonography-CT/MRI fusion guidance for percutaneous ablation of inconspicuous, small liver tumors: improving feasibility and therapeutic outcome. Cancer Imaging. 2024 Jan 3;24(1):4. doi: 10.1186/s40644-023-00650-y. PMID 38172949